CLINICAL TRIAL: NCT04099381
Title: Protocol for Evaluating the Safety and Efficacy of Transfusion of Umbilical Cord Blood in Patients With a Diagnosis of Autism Spectrum Disorder Depending on the Degree of Tissue Compatibility of the Donor and the Recipient
Brief Title: Safety and Efficacy of the Transfusion of UCB in Patients With an ASD Depending on the Degree of HLA Compatibility.
Acronym: ASD-HLA2019
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Collaborators: INBIO, LLC (Unknown)
Responsible Party: Principal Investigator, Volchkov Stanislav, Deputy director, Quality assurance director, State-Financed Health Facility "Samara Regional Medical Center Dinasty"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASD-HLA2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Autism, ASD, Cord blood, HLA
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is prospective, non-randomized (open-label) with control group study. In total, the study will involve 150 patients in three groups. The first and second groups will receive transfusions of umbilical cord blood hematopoietic cells, with varying degrees of selection for the genes of the HLA system. The third group will be the control group. In the control group, 50 patients with similar pathology will be examined, comparable in age, sex and degree of disorder of the type of "para-copies" against the background of standard therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Low HLA compatibility (Experimental): ASD CB-MNC infusion from different donors and standard therapy. CBU with 3 or less HLA compatibility degree in A, B, DRB1 loci will be used.
  Interventions: Biological: ASD CB-MNC infusion low level HLA compatibility.
- Group 2 High HLA compatibility (Experimental): ASD CB-MNC infusion from different donors and standard therapy. CBU with 3 or more HLA compatibility degree in A, B, DRB1 loci will be used.
  Interventions: Biological: ASD CB-MNC infusion high level HLA compatibility.
- Group 3 Control (Other): Patients with standard therapy as a control group.
  Interventions: Other: Standard therapy.

INTERVENTIONS:
Biological: ASD CB-MNC infusion low level HLA compatibility. — CB-MNC infusion from different donors. One dose consists of 2-15х10^7 cells per 1 kg of patient weight for each infusion. The protocol includes 2 infusions with an interval of 6-x months. HLA compatibility of the cord blood is 3 or fewer by A, B, DRB1 loci.
  Arms: Group 1 Low HLA compatibility
Biological: ASD CB-MNC infusion high level HLA compatibility. — CB-MNC infusion from different donors. One dose consists of 2-15х10^7 cells per 1 kg of patient weight for each infusion. The protocol includes 2 infusions with an interval of 6-x months. HLA compatibility of the cord blood is 4 or more by A, B, DRB1 loci.
  Arms: Group 2 High HLA compatibility
Other: Standard therapy. — The standard therapy can include drugs, special psychology training etc.
  Arms: Group 3 Control

SUMMARY:
Autism is one of those disorders in Autism spectrum disorders (ASD), which characterized by social interaction abnormalities, impaired verbal and non-verbal communication, and repetitive, obsessive behavior, while the therapeutic effect of current treatments remains limited progress.

The possible reason for ASD is neural hypoperfusion and immune dysregulation. The Human Umbilical Cord Blood Mononuclear Cells (hUCB-MNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy. In this study, the safety and efficacy of hUCB-MNCs infusion will be evaluated in patients with Autism with regarding to HLA compatibility.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are heterogeneous neuro-developed disorders. Autism is the most common disorder of the diseases characterized by dysfunctions in response to social interaction and communication, as well as the presence of repetitive and stereotyped behaviors. Recent reports of a sharp increase in the number of children with autism. The exact etiology of autism remains unclear. Compliance, the definition of effective treatments for autism is particularly difficult.

Although it has been understood, it can be a question of immune dysregulation. Examination of the inflammatory cytokines, dysfunction of the immune system and the immune system. The Human Umbilical Cord Blood Mononuclear Cells (hUCB-MNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy. Our study suggest that infusion of cord blood mononuclear cells will affect Autism.

This protocol was developed on the basis of the results of the previously approved protocol of the center NCT03786744 (Transfusion of allogeneic cord blood samples in patients with autism spectrum disorders), which showed high efficiency in the rehabilitation of patients. The present protocol is intended for revealing the dependence of the clinical effect on the degree of tissue compatibility of umbilical cord blood samples and the recipient.

ELIGIBILITY:
Patient selection criteria (indications for this type of treatment):

* Patient's age from 4 to 14 years;
* Diagnosis: autistic spectrum disorder;
* The severity of the disease on the ATEC scale of at least 16 points;
* The presence of a compatible allogeneic sample suitable for infusion;
* Parental consent (official guardians).

Patient exclusion criteria (contraindications for this type of treatment):

* The patient's age under 4 years, after 14 years;
* The presence of the following diseases in the history: heart failure at the stage of decompensation, stroke in the history of less than 1 year ago, anemia and other blood diseases;
* Decompensation for chronic and endocrinological diseases;
* Acute viral and bacterial infections during the acute clinical phase of the disease;
* HIV infection, hepatitis B and C;
* Cancer, chemotherapy, and history of cancer;
* Tuberculosis;
* Severe form of intellectual disability as a concomitant disease (diagnosis can be ignored, according to the decision of the Medical Committee of the Center);
* Fragile X chromosome syndrome;
* Epileptic seizures with or without medication in the last 6 months before inclusion in the protocol.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with non-serious and serious adverse events. | baseline, change from baseline at 12 month
  Safety assessment. Adverse events rate will be assessed in all patients.
The Childhood Autism Rating Scale (CARS2). | baseline, change from baseline at 6,12 month
  Rating for behavior, characteristics, and abilities against the expected developmental growth. Will be assessed fifteen items, including: relationship to people; imitation; emotional response; body; object use; adaptation to change; visual response; listening response; taste-smell-touch response and use; fear and nervousness; verbal communication; non-verbal communication; activity level; level and consistency of intellectual response; general impressions. Total score will be assessed. Scores range form 15 to 60 with 30 being the cutoff rate for a diagnosis of mild autism. Scores 30-37 indicate mild to moderate autism, while scores between 38 and 60 are characterized as severe autism.
Autism Treatment Evaluation Checklist (ATEC). | baseline, change from baseline every month (total 12 evaluations)
  Will be assessed: I. Speech/Language Communication (14 items); II. Sociability (20 items); III. Sensory/ Cognitive Awareness (18 items); and IV. Health/Physical/Behavior (25 items).

SECONDARY OUTCOMES:
Evaluation of the survival of donor cells in the host body without immune responses | baseline, change from baseline at 6 month
  Evaluation of the survival of donor cells in the host body to determine the safety and duration of the cellular component. To do this, before the first injection of the cells, a sample of the patient's blood and a donor cord blood sample will be taken. 6 months after the first injection of the cells, immediately before the second injection, the patient's blood will be re-taken to conduct a study on chimerism. The obtained data will allow assessing the survival degree of donor material. The definition of chimerism is carried out by fragment analysis. For analysis, blood samples of the biomaterial will be collected from the patient before the cells are injected and 6 months after the injection.
The correlation of the concentration of T-regulatory cells (CD4/CD25/FoxP3) in the sample of umbilical cord blood and the treatment effectiveness degree | At 1, at 6 months (At first and second infusion)
  A correlation between the concentration of cells of the monocyte-macrophage series (CD4/CD25/FoxP3) and the degree of recovery of neurological functions. This information will be used to assess treatment effectiveness. The assessment of a cord blood sample will be carried out on a flow cytometer immediately before the injection of the cells or in the next 12 hours.
The correlation of the concentration of T-regulatory cells (CD4/CD25/FoxP3) in the patient depending on the severity of the disease. | At 1, at 6 months (At first and second infusion)
  A correlation between the concentration of T regulatory cells (CD4/CD25/FoxP3) and the severity of the disease. This information will be used to assess treatment effectiveness. The assessment of a cord blood sample will be carried out on a flow cytometer immediately before the first injection of the cells, and before the second injection of the cells.
The correlation of the concentration of CD34+ cells in the cord blood sample and the treatment effectiveness degree | At 1, at 6 months (At first and second infusion)
  CD34+ cells are precursors of hematopoiesis and endothelium. Studies show that CD34+ cells, when injected into an ischemic lesion zone, exert protective properties on the affected cells, stimulate angiogenesis, and are involved in reducing inflammatory reactions. In this study, we plan to find a correlation between the concentration of the introduction of CD34+ cells and treatment effectiveness. The assessment of a cord blood sample will be carried out on a flow cytometer immediately before the injection of the cells or in the next 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: STANISLAV VOLCHKOV, MD, PhD, Principal Investigator — Medical Centre Dinasty
Locations (1):
- Medical Centre Dinasty, Samara, Russia